CLINICAL TRIAL: NCT05731258
Title: Clinical Observational Study of Postoperative Adjuvant Treatment of Breast Cancer With Liposomal Doxorubicin Regimen
Brief Title: Observational of Adjuvant Treatment of Breast Cancer With Liposomal Doxorubicin Regimen
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0239
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Liposomal Doxorubicin; Efficacy; Safety; Postoperative Adjuvant Treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Liposomal doxorubicin containing regimen — Liposomal doxorubicin hydrochloride (PLD) 30-40mg/m2 D1 + other drugs (decided by investigators); All patients were treated with 4 cycles.

SUMMARY:
The goal of this observational study aims to observe and evaluate the efficacy and safety of a liposomal doxorubicin containing regimen in the postoperative adjuvant treatment of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18-75 years;
2. Primary breast cancer diagnosed histopathologically;
3. Adjuvant chemotherapy regimens include liposomal doxorubicin;
4. ECoG PS score: 0-1 points;
5. Left ventricular ejection fraction (LVEF) ≥ 55%;
6. Estimated survival ≥ 6 months;
7. Major organ function is normal, i.e. meets the following criteria:

   ① And white blood cells ≥ 4.0 × 10 9 / L, neutrophil count (ANC) ≥ 1.5 × 10 9 /L；② Platelets ≥ 100 × 10 9 /L；③ And hemoglobin ≥ 10 g / dl; ④ Serum creatinine ≤ 1.5 × ⑤ the upper limit of normal (ULN) Mmol / L and aspartate transaminase (AST) ≤ 2.5

   × ULN；⑥ Alanine transaminase (ALT) ≤ 2.5 × ULN；⑦ Total bilirubin ≤ 1.5 × ULN；⑧ Serum creatinine ≤ 1.5 × ULN；
8. Subjects voluntarily join this study, sign the informed consent form, have good compliance and cooperate with follow-up.

Exclusion Criteria:

1. Pregnant, lactating patients;
2. Breast cancer has been found to have distant metastasis;
3. Those with peripheral nervous system disorders caused by the disease or with a history of significant mental disorders and central nervous system disorders;
4. Those with severe infection or active peptic ulcer requiring treatment;
5. Allergic to chemotherapy drugs;
6. Cancer free period less than 5 years except for cured basal cell carcinoma of the skin and cured carcinoma in situ of the cervix;
7. Severe liver disease (e.g., cirrhosis, etc.), renal disease, respiratory disease, or uncontrolled diabetes;
8. Patients who are participating in other clinical trials or within a month.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early breast cancer patients who required four cycles of chemotherapy after curative resection of breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Cardiac safety | 10 years
  Cardiac ejection fraction

SECONDARY OUTCOMES:
Overall survival | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliate Hospital of Zhejiang University, Hangzhou, Zhejiang, China